CLINICAL TRIAL: NCT02743299
Title: Investigation of a Novel Turbine-driven Ventilator for Use in Cardiopulmonary Resuscitation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Scott Allen, Anesthesiologist, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00063298
Record Dates: First submitted 2016-04-01; First posted 2016-04-19 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Arrest; Hyperventilation
MeSH Terms: conditions — Heart Arrest; Hyperventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPR simulation (Experimental): CPR simulation with and without ventilator
  Interventions: Device: Handivent Ventilator

INTERVENTIONS:
Device: Handivent Ventilator — CPR with use of a turbine-driven ventilator (Handivent)

SUMMARY:
The objective of this study is to determine whether healthcare professionals trained in CPR can deliver more effective ventilations during CPR using the Handivent, a novel turbine-driven ventilator as compared to bag-valve-mask ventilations, using a manikin model. The investigators believe the Handivent will deliver a more accurate respiratory rate and tidal volume, with lower intrathoracic pressure during CPR.

DETAILED DESCRIPTION:
Previous studies have shown that increased respiratory rate during CPR inversely correlates with blood pressure. Higher respiratory rates increase intrathoracic pressure, which in turn decreases venous return to the heart.

In one previous study, the authors looked at 3 groups of 7 pigs, ventilated at 12 (100% O2), 30 (100%), and 30 (5% CO2, 95% 02) breaths per minute during cardiac arrest, and showed increased mortality with increasing respiratory rate. Survival rates were 6/7, 1/7, and 1/7 respectively. The results of this study led to changing the CPR guidelines in 2005 to include fewer ventilations.

The authors also observed 13 cases of CPR in the field and noted EMS personnel delivered breaths at an average of 32 bpm.

In 2012, a similar study to the current study under proposal compared a pressure-limited, pneumatically driven ventilator to bag-valve-mask in simulated CPR, using medical student volunteers. That study did not show a significant difference in tidal volumes; however, they did not record respiratory rates or mean intrathoracic pressures. Furthermore, that ventilator was pneumatically -driven and pressure limited, whereas the ventilator we propose to study is turbine-driven and can be volume/time triggered.

ELIGIBILITY:
Inclusion Criteria:

* ACLS- certified healthcare professional

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | RR will be the average RR during the CPR simulation, which is 8-minutes in duration.
  The study will measure the respiratory rate delivered during the 8-minute CPR scenario

SECONDARY OUTCOMES:
Tidal volume | Average Vt during CPR simulation, which is 8 minutes in duration
  The study will measure the tidal volume delivered during the 8-minute CPR scenario
Peak Inspiratory pressure | Average PIP delivered during CPR simulation, which is 8 minutes in duration.
  the study will measure the peak inspiratory pressure delivered during the 8-minute CPR scenario

CONTACTS AND LOCATIONS:
Overall Officials: Scott Allen, MD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen SG, Brewer L, Gillis ES, Pace NL, Sakata DJ, Orr JA. A Turbine-Driven Ventilator Improves Adherence to Advanced Cardiac Life Support Guidelines During a Cardiopulmonary Resuscitation Simulation. Respir Care. 2017 Sep;62(9):1166-1170. doi: 10.4187/respcare.05368. Epub 2017 Aug 14. PMID 28807986